CLINICAL TRIAL: NCT02674529
Title: Study of Neural Responses Induced by Simulated Antidepressants
Brief Title: Study of Neural Responses Induced by Antidepressant Effects
Acronym: SONRISA
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Marta Peciña, MD PhD (Other)
Responsible Party: Sponsor-Investigator, Marta Peciña, MD PhD, Assistant Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STUDY19070392/PRO16050131
Record Dates: First submitted 2016-01-22; First posted 2016-02-04 (Estimated); Results first posted 2022-11-03 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-10

CONDITIONS: Major Depressive Disorder
Keywords: Depression; Neuroimaging biomarkers; MDD; Neurofeedback
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Escitalopram

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Antidepressant Treatment (Active Comparator): 20mg of escitalopram will be taken over an 8-week period, starting with 10mg for the first week.
  Interventions: Drug: Escitalopram; Behavioral: Real-time Neurofeedback fMRI task pre- and post-RCT
- Placebo (Placebo Comparator): A placebo pill will be taken over an 8-week period.
  Interventions: Drug: Placebo; Behavioral: Real-time Neurofeedback fMRI task pre- and post-RCT

INTERVENTIONS:
Drug: Escitalopram — Selective Serotonin Reuptake Inhibitor (SSRI)
  Other Names: Lexapro
  Arms: Antidepressant Treatment
Drug: Placebo — Placebo
  Arms: Placebo
Behavioral: Real-time Neurofeedback fMRI task pre- and post-RCT — Placebo experiment during an fMRI scanning session

SUMMARY:
The proposed work aims to examine the neural changes associated with fast-acting antidepressant treatments in order to develop imaging-based biomarkers of treatment response for depression.

DETAILED DESCRIPTION:
Over the past decade, neuroimaging tools have rapidly advanced the field of neural biomarkers of treatment response in depression. Still, despite obvious scientific progress in this field, the ability to implement neuroimaging biomarkers of antidepressant treatment response in clinical trial settings is lacking. In order to objectively assess the neural bases of treatment response in depression, the investigators will use a "Real-time Neurofeedback fMRI task", specifically designed to record and modulate mood improvement by providing neurofeedback in the context of the administration of an antidepressant treatment. In a pilot study, positive neurofeedback during the administration of the drug was associated with significant acute mood improvement and increased blood oxygen level dependent (BOLD) responses in the rostral anterior cingulate cortex (rACC), a common neural target of antidepressant treatments. The central hypothesis is that antidepressant effects in depression are mediated by increased neural activity in the rACC (AIM1), which can be used in clinical trials of antidepressant treatment to predict antidepressant effects (AIM 2) and assess the effect of antidepressant treatment on antidepressant-induced rACC neural responses (AIM 3). The results obtained from this project are expected to have an important impact on our ability to understand the cognitive and neural mechanisms implicated in antidepressant treatment responses in patients with depression, as well as on the ability to implement neuroimaging biomarkers of treatment response in the clinical trial settings.

ELIGIBILITY:
Inclusion Criteria:

* A man or woman age of 18 or older.
* Currently experiencing a depressive episode as part of Major Depressive Disorder.
* Able to tolerate lying still on your back for 60 minutes at a time.
* Have had no more than one failed antidepressant trial of adequate dose and duration.
* Have been antidepressant medication-free for at least 21 days prior to collection of imaging data (5 weeks for fluoxetine)

Exclusion Criteria:

* Are currently taking any psychiatric medication, or any potentially augmenting or sedative drugs.
* Have a history of inadequate response/tolerability to escitalopram; or history of resistant depression
* Pregnant or breastfeeding or plan to become pregnant over the duration of the study.
* Have a history (lifetime) of psychotic depressive, schizophrenic, bipolar, schizoaffective, or other Axis I psychotic disorders.
* Meet criteria for substance dependence in the last 6 months, except nicotine, or substance abuse in the last 2 months.
* Have a medical condition that contradicts treatment with escitalopram.
* Are currently receiving psychotherapy or any other treatment for your depression.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2021-05 (Actual); Study Completion 2021-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marta Pecina, MD, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- WPIC, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
The study will follow NIMH schedule for data sharing for clinical trials. The schedule allows for descriptive data to be submitted - but not shared - ongoing and results associated with a finding - both positive and negative - to be submitted prior to the communication of a result. Once a result is communicated, either through publication and/or on the NDCT website the data specifically defined to the clinical trial will then be shared.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Six participants were excluded after enrollment for the following reasons: leaving the study site without informing study team, asking for extra-time to consider the study, feeling uncomfortable in the fMRI and asking to exit the scanner, testing positive for pregnancy tests, feeling indecisive, and not responding to contact attempts.
Period: Overall Study
Arm/Group | Antidepressant Treatment | Placebo
Started | 25 | 29
Completed | 22 | 24
Not Completed | 3 | 5
Not completed — Lost to Follow-up | 1 | 2
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Physician Decision | 0 | 1
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Antidepressant Treatment | Placebo | Total
Number analyzed (Participants) | 25 | 29 | 54
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 25 | 29 | 54
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.44 (6.33) | 23.45 (5.65) | 24.18 (5.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 26 | 46
  Male | 5 | 3 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 23 | 29 | 52
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 6 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 8 | 10
  White | 14 | 15 | 29
  More than one race | 5 | 0 | 5
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 25 | 29 | 54

OUTCOME MEASURES:

1. Primary Outcome: Change in Montgomery-Åsberg Depression Rating Scale (MADRS) Scores
Description: The Montgomery-Åsberg Depression Rating Scale (MADRS) is a ten-item diagnostic questionnaire which psychiatrists use to measure the severity of depressive episodes in patients with mood disorders. It was designed in 1979 by British and Swedish researchers as an adjunct to the Hamilton Rating Scale for Depression (HAMD) which would be more sensitive to the changes brought on by antidepressants and other forms of treatment than the Hamilton Scale was.[2] There is, however, a high degree of statistical correlation between scores on the two measures.
Time Frame: baseline and week 8
Population: Scores can range from 0-60, with higher scores meaning greater the depression severity. The greater the change in MADRS scores from baseline, the better the outcome. 46 participants were analyzed, with 8 participants lost to follow up.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Changes in MADRS Scores From Baseline to Week 8 Within the Antidepressant Treatment Arm: 20mg of escitalopram will be taken over an 8-week period, starting with 10mg for the first week.
  Escitalopram: Selective Serotonin Reuptake Inhibitor (SSRI)
- Changes in MADRS Scores From Baseline to Week 8 Within the Placebo Arm: A placebo pill will be taken over an 8-week period.
  Placebo: Placebo
Arm/Group | Changes in MADRS Scores From Baseline to Week 8 Within the Antidepressant Treatment Arm | Changes in MADRS Scores From Baseline to Week 8 Within the Placebo Arm
Number analyzed (Participants) | 22 | 24
score on a scale | 11 (9) | 12 (9)
Statistical Analysis 1: Comparison: Changes in MADRS Scores From Baseline to Week 8 Within the Antidepressant Treatment Arm vs Changes in MADRS Scores From Baseline to Week 8 Within the Placebo Arm; Test type: Other — This was a mechanistic trial and non-inferiority or equivalence analysis were not performed; p = 0.58, Regression, Linear; Drug (antidepressant vs. placebo) prediction of changes in mood as measured by the MADRS scores; regression coefficient = -1.29864, Standard Error of Mean 2.3
Statistical Analysis 2: Comparison: Changes in MADRS Scores From Baseline to Week 8 Within the Antidepressant Treatment Arm vs Changes in MADRS Scores From Baseline to Week 8 Within the Placebo Arm; Test type: Other; p = 0.05, Correlation; Change in MADRS after 8 weeks correlation with brain responses during the baseline fMRI task; r = 0.02

2. Secondary Outcome: Change in Quick Inventory of Depressive Symptomatology (QIDS) Scores
Description: The Quick Inventory of Depressive Symptomatology (QIDS) is a 16-item, self-reported measure of depression that ranges from 1 (no depression) to 27 (very severe depression).
Time Frame: baseline and 8 weeks
Population: Scores can range from 0-27, with higher scores meaning greater the depression severity. The greater the change in QIDS scores from baseline to week 8, the better the outcome. 46 participants were analyzed, with 8 participants lost to follow up.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Changes in QIDS Scores From Baseline to Week 8 Within the Antidepressant Treatment Arm: 20mg of escitalopram will be taken over an 8-week period, starting with 10mg for the first week.
  Escitalopram: Selective Serotonin Reuptake Inhibitor (SSRI)
- Changes in QIDS Scores From Baseline to Week 8 Within the Placebo Arm: A placebo pill will be taken over an 8-week period.
  Placebo: Placebo
Arm/Group | Changes in QIDS Scores From Baseline to Week 8 Within the Antidepressant Treatment Arm | Changes in QIDS Scores From Baseline to Week 8 Within the Placebo Arm
Number analyzed (Participants) | 22 | 24
score on a scale | 6.82 (6.01) | 5.54 (5.45)
Statistical Analysis 1: Comparison: Changes in QIDS Scores From Baseline to Week 8 Within the Antidepressant Treatment Arm vs Changes in QIDS Scores From Baseline to Week 8 Within the Placebo Arm; Test type: Other — This is a mechanistic trial, we did not perform non-inferiority or equivalence analysis; p = 0.8, Regression, Linear; regression coefficient = -1.4328918, Standard Deviation 1.4

3. Secondary Outcome: Neural Responses During the Sham Neurofeedback fMRI Task.
Description: Voxel-wise BOLD changes during the expectancy condition of the Sham Neurofeedback fMRI task.
Time Frame: Baseline
Measure: Mean (Inter-Quartile Range); unit: BOLD signal change
Groups:
- Baseline fMRI Measures: The primary objective is to define the neural correlates of placebo response in MDD.
Arm/Group | Baseline fMRI Measures
Number analyzed (Participants) | 54
BOLD signal change | 1.1 [0.47 to 1.61]
Statistical Analysis 1: Comparison: Baseline fMRI Measures; At the group-level, a random-effects analysis determines the main effects of the regressors of interest (e.g., high vs. low expectancy) resulting in statistical parametric maps (t or F statistics). To control for potential confounders, sex and depression severity will be entered as covariates in statistical models; Test type: Other; p < 0.05, t-test, 2 sided — The resulting voxel-wise parametric maps are thresholded with height and extent values generated by Monte Carlo simulations with 3dClustSim to protect against overall type I error at p < 0.05

ADVERSE EVENTS:
Time Frame: Eight weeks.
Arm/Group | Antidepressant Treatment | Placebo
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/29
Other Adverse Events (participants affected / at risk) | 22/25 | 18/29
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Antidepressant Treatment (N=25) | Placebo (N=29)
Appetite Disturbances (Gastrointestinal disorders) | 6 (8) | 1 (1)
Gastrointestinal Discomfort (Gastrointestinal disorders) | 3 (6) | 2 (2)
Nausea (Gastrointestinal disorders) | 6 (9) | 3 (7)
Weight Loss (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 5 (5) | 2 (2)
Vivid Dreams/Nightmares (Nervous system disorders) | 2 (4) | 0 (0)
Headache (Nervous system disorders) | 3 (3) | 2 (3)
Worsening of Depressive Symptoms (Nervous system disorders) | 2 (3) | 1 (1)
Anxiety (Nervous system disorders) | 2 (2) | 3 (6)
Distractibility (Nervous system disorders) | 0 (0) | 1 (1)
Hypomania (Nervous system disorders) | 0 (0) | 1 (1)
Insomnia (General disorders) | 3 (4) | 5 (5)
Fatigue (General disorders) | 12 (31) | 5 (6)
Yawning (General disorders) | 2 (2) | 0 (0)
Dry Mouth (General disorders) | 1 (6) | 0 (0)
Increased Thirst (General disorders) | 2 (7) | 1 (3)
Palpitations/Increased Heart Rate (General disorders) | 1 (4) | 1 (1)
Sweating (General disorders) | 1 (1) | 0 (0)
Sexual Dysfunction (General disorders) | 2 (6) | 0 (0)
Urinary Urgency (General disorders) | 0 (0) | 2 (5)
Leg Pain (Social circumstances) | 1 (1) | 0 (0)
Cold/Sore Throat (Social circumstances) | 1 (1) | 1 (1)
Broken Wrist (Social circumstances) | 1 (2) | 0 (0)
Ovarian Cyst Rupture (Social circumstances) | 1 (1) | 0 (0)
Food Poisoning (Social circumstances) | 0 (0) | 1 (1)
Vision Issues (Social circumstances) | 0 (0) | 1 (2)
Urinary Tract Infection (Social circumstances) | 0 (0) | 1 (1)
Gonorrhea (Social circumstances) | 0 (0) | 1 (2)
COVID-19 (Social circumstances) | 0 (0) | 1 (2)
Teeth Grinding/Jaw Clenching (Social circumstances) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-29): https://cdn.clinicaltrials.gov/large-docs/29/NCT02674529/Prot_SAP_000.pdf